CLINICAL TRIAL: NCT04734067
Title: Exploration of Predictive Markers and Establishment of Predictive Models for Checkpoint Inhibitor Pneumonitis in Combination With Imaging in Immune Checkpoint Inhibitor Therapy
Brief Title: Exploration of the Predictive Marker and Establishment of Predictive Models of Checkpoint Inhibitor Pneumonitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Tang-Du Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Henan Cancer Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2021LSK-001
Record Dates: First submitted 2021-01-12; First posted 2021-02-02 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Pneumonia, Interstitial
Keywords: immune checkpoint inhibitors; predictive marker; predictive model; immunotherapy
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fasting venous blood was drawn from patients who first received immune checkpoint inhibitors therapy before baseline and before cycle 3，5...2n+1.Then the blood samples were centrifuged and frozen in a refrigerator at -80℃ for later mass spectrometry analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational group: Patients receiving ICIs for the first time
  Interventions: Other: Immune checkpoint inhibitors(ICIs) therapy

INTERVENTIONS:
Other: Immune checkpoint inhibitors(ICIs) therapy — Patients with malignant tumors who first received ICIs

SUMMARY:
This is a prospective, multicenter observational study to explore the predictive factors of checkpoint inhibitor pneumonitis (CIP) and to establish predictive models by combining imaging information for IRP. The imaging type of CIP, the pathological type, various inflammatory cytokines and tumor proportion score(TPS) of PD-L1 expression level, etc. will be paid more attention.

DETAILED DESCRIPTION:
Prospective dual-arm, multicenter observational study to explore the predictive factors of checkpoint inhibitor pneumonitis (CIP) and to establish predictive models by combining imaging information.Patients will receive work-up, treatment and follow-up exclusively as routinely done except monitoring and evaluation of CIP. Necessary tests will be required, such as lung function tests, lymphocyte subsets, and thin-section CT of the chest during evaluation of the disease.This study mainly included patients with malignant tumor who received immune checkpoint inhibitors for the first time.Fasting venous blood was taken before treatment and before cycle 3,5...2n+1 of treatment. Then the blood samples were centrifuged and frozen in a refrigerator at -80℃ for later mass spectrometry analysis. IrAEs of patients was strictly recorded according to CommonTerminology Criteria Adverse Events V4.0 (CTCAE V4.0). The main objective was to explore the relationship between various indicators and the occurrence of CIP, including pulmonary ventilation and diffusion function at baseline, C-reative protein(CRP), cytokines, interleukin-6(IL-6), CD4+ T lymphocyte count and percentage, CD8+ T lymphocyte count and percentage, NK cell count and percentage, total T lymphocyte count and percentage, neutrophil counts and percentages, eosinophilic cell count and percentage, white blood cell count, blood platelet count, serum albumin(ALB), alanine aminotransferase(ALT), aspartate aminotransferase (AST), γ-glutamyl transpeptadase（γ-GGT), body mass index (BMI), serum procalcitonin(PCT), smoking index and various inflammatory cytokines.

Primary study endpoints: The predictive factors and the predictive models of CIP.

Secondary study endpoints: The incidence and clinical characteristics of CIP.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* Obtain written informed consent and any locally required authorization from the patient or his/her legal representative prior to the commencement of any study protocol related procedures, including screening assessments;
* Patients with malignant tumors confirmed by histology or cytology can be treated with ICIs after evaluation by a professional oncologist, with no restriction on cancer type or stage;
* Life expectancy on day 1 ≥12 weeks;
* When selected, the Eastern Cooperative Oncology Group (ECOG) physical status score was 0-2;
* No previous use of immunotherapy；
* No prior exposure to immune-mediated therapy;
* Have sufficient viscera function and bone marrow function;
* Evidence of postmenopausal status in women, or negative urine or serum pregnancy tests in premenopausal women.

Exclusion Criteria:

* The target lesion had received immune-related treatment or immune-mediated treatment before;
* Patients with clinically confirmed moderate to severe pulmonary interstitial fibrosis before taking ICIs;
* Major surgical procedures were performed within 28 days of the first medication;
* History of allograft transplantation;
* Active or previously documented autoimmune or inflammatory diseases or other contraindications for immunotherapy;
* Uncontrolled serious complications such as infection and acute cardio-cerebrovascular disease;
* The presence of another primary malignancy;
* anaphylaxis or hypersensitivity to immunotherapy or chemotherapy;
* Decompensation of viscera and low bone marrow function and hematopoietic function；
* Pregnant or lactating female patients;
* Expected survival time < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant tumor receiving immune checkpoint inhibitors for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2021-08-20 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The change of C reactive protein(CRP); mg/L | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  CRP level in the serum.
Interleukin-6(IL-6); Pg/ml | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  IL-6 level in the serum.
CD4+ T lymphocyte; /uL | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The absolute and relative counts of CD4+ T lymphocyte in whole blood.
CD4+ T lymphocyte; percent | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  Percentage of CD4+ T lymphocyte in whole blood.
CD8+ T lymphocyte; /uL | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The absolute and relative counts of CD8+ T lymphocyte in whole blood.
CD8+ T lymphocyte; percent | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  Percentage of CD8+ T lymphocyte in whole blood.
NK cell; /uL | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The absolute and relative counts of NK cell in whole blood.
NK cell; percent | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  Percentage of NK cell in whole blood.
White blood cell count; 10^9/L | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The white blood cell count in whole blood.
Lymphocyte count; 10^9/L | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The absolute and relative counts of total lymphocyte count in whole blood.
Lymphocyte count; percent | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  Percentage of total lymphocyte count in whole blood.
Eosinophils count; 10^9/L | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The absolute and relative counts of eosinophils count in whole blood.
Eosinophils count; percent | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  Percentage of eosinophils count in whole blood.
Blood platelet count; 10^9/L | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The blood platelet count in whole blood.
Alanine aminotransferase(ALT); U/L | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The ALT level in the serum.
Aspartate aminotransferase (AST); U/L | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The AST level in the serum.
Serum albumin; g/L | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The albumin level in the serum.
γ-glutamyl transpeptadase（γ-GGT); U/L | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The γ-GGT level in the serum.
Smoking index | At baseline
  The average root number per day multiplied by smoking years of smoking, that is, smoking index.
Body mass index (BMI); kg/m^2 | At baseline
  The body's weight(Kg) divided by the square of your height(m), that is, body mass index.
Serum procalcitonin(PCT); ng/ml | Before Cycle 1,3, 5, 7 and 2n+1(each cycle is 21 days) and through study completion, an average of 6 months.
  The PCT level in the serum.
Forced vital capacity(FVC); L | Before Cycle 1.
  The maximum amount of air that can be exhaled as soon as possible after the maximum inhalation. FVC was used to evaluate pulmonary ventilation function.
Forced the first second of expiratory volume (FEV1); L | Before Cycle 1.
  the first second of exhalation during the maximum exhalation after the maximum deep inhalation. FEV1 was used to evaluate pulmonary ventilation function.
FEV1/FVC; percent | Before Cycle 1.
  FEV1 accounts for the percentage of FVC. FEV1/FVC was used to evaluate pulmonary ventilation function.
Maximal mid-expiratory flow(MMEF); L/s | Before Cycle 1.
  The average flow rate with forced exhalation of 25% to 75% of lung capacity. FEV1/FVC was used to evaluate pulmonary ventilation function.
Fractional exhaled nitric oxide (FeNO) measurement；ppb | Before Cycle 1.
  FeNO measurement quantified the amount of nitric oxide (NO) in one's exhaled breath, which was used to evaluate pulmonary diffusion function.

SECONDARY OUTCOMES:
The incidence of IRP; percent | Up to 36 months
  The incidence of IRP in the general population receiving ICIs

CONTACTS AND LOCATIONS:
Overall Officials: Hui Guo, PH.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: Undecided